CLINICAL TRIAL: NCT05002673
Title: Determination of the Effect of Two Different Methods of Dental Anaesthesia on Pain Level in Paediatric Patients: A Cross-over, Randomised Trial
Brief Title: Dental Anaesthesia Affects Pain Level
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karadeniz Technical University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Nagehan Yilmaz, Assistant Prof, Karadeniz Technical University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Karadeniz
Record Dates: First submitted 2021-07-16; First posted 2021-08-12 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2021-08

CONDITIONS: Dental Anxiety; Anesthesia, Local

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SLEEPERONE (Experimental)
  Interventions: Device: DENTAL LOCAL ANESTHESİA
- COMFORTIN (Experimental)
  Interventions: Device: DENTAL LOCAL ANESTHESİA

INTERVENTIONS:
Device: DENTAL LOCAL ANESTHESİA — doing local and topical anesthesia with two different device

SUMMARY:
Background: Needles are the most feared tools, making anaesthetic injection a worrying practice.

Aim: To compare intraosseous (IOA) and needle-free dental anaesthesia (NFA) methods that painless anaesthesia.

Design: Twenty patients aged 8-10 years were included in this cross-over study. To determine the anxiety levels and pain experienced by the patients, visual and behavior scales were used. The pulse rate (PR) and opiorphin levels (OL) determined. The Friedman and Wilcoxon signed-rank tests were used. p<0.05 was considered significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 8-10 years,
* systemically healthy,
* had undergone dental treatment (except for extraction) previously but with at least 1 week passed since then
* were compatible enough to undergo therapy in the clinic in a sitting position,
* had infection between the roots with a rate over 1/3, had 2/3 root formation,
* had been indicated for extraction of the maxillary primary molar teeth (55/65 No. teeth),
* did not have acute and/or subacute infection of the related or other teeth or mouth and surrounding tissues

Exclusion Criteria:

* who scored above 41 in the state anxiety subscale and above 44 in the trait anxiety subscale of the Spielberger State-Trait Anxiety Scale (SSAS-SAAS)
* not meeting the inclusion criteria

Ages: 8 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Score of scales (wong baker faces pain rating scale) | one year
  (0-10) (0= no hurt, 10= hurts worst)
Score of scales (face, legs, activity, cry, consolability) | one year
  (0-10) (0= relaxed, 10=severe discomfort)
Score of scales (frankl behavior rating scale) | one year
  (1-4) (1= definitely negative, 4=definitely positive)
heart rate (pulse oximeter) | one year
level of opiorphin (from saliva samples) | one year

CONTACTS AND LOCATIONS:
Locations (1):
- Nagehan Yılmaz, Trabzon, None Selected, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No